CLINICAL TRIAL: NCT06992050
Title: Comparative Evaluation of the Thermal Protection Provided by Submarine Rescue Suits: Half Suit Versus Full Suit
Status: Completed | Type: Observational
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Dror Ofir, PHD, Medical Corps, Israel Defense Force
Other Study IDs: 1895 - 2018
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cold Exposure, Hypothermia, Thermal Insulation, Immersion Suits, Submarine Evacuation
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Full Suit Group: Participants wearing full-body Submarine Escape Immersion Equipment (SEIE) suits
  Interventions: Device: Submariner suit
- Half Suit Group: Participants wearing half-body Submarine Escape Immersion Equipment (SEIE) suits
  Interventions: Device: Submariner suit

INTERVENTIONS:
Device: Submariner suit — Participants wearing full-body Submarine Escape Immersion Equipment (SEIE) suits

SUMMARY:
This study evaluated the thermal and functional performance of full-body versus half-body Submarine Escape Immersion Equipment (SEIE) suits during cold water immersion (~16.5°C) and raft sitting. Twenty submariners were divided into two groups.

DETAILED DESCRIPTION:
This study investigates the performance of full-body versus half-body Submarine Escape Immersion Equipment (SEIE) suits under conditions simulating submarine emergencies in cold water (~16.5°C). In such scenarios, rapid evacuation and prolonged exposure to cold water pose significant risks of hypothermia and impaired physical function. The aim was to assess and compare the thermal insulation and motor performance effects of both suit designs during water immersion and raft sitting.

Twenty healthy active-duty submariners (age 22 ± 1 years) participated, divided evenly into two groups (full suit vs. half suit). Core temperature was monitored using ingestible sensors, and subjective cold sensation was assessed regularly throughout immersion and raft sitting. Additional outcome measures included fine motor dexterity (assembling shackles) and handgrip strength, recorded before and after exposure.

The experimental protocol involved one session per participant. Anthropometric data were collected, and subjects underwent a controlled immersion and raft sitting protocol using calibrated thermal equipment. Motor function tasks were standardized and repeated to control for learning effects. Statistical analysis included non-parametric repeated measures tests with appropriate corrections for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

Healthy active-duty submariners

Male participants aged 20-25 years

No history of cardiovascular, respiratory, or neurological disorders

Not acclimatized to cold environments or cold water exposure

Provided written informed consent

Medically cleared for cold water immersion by a physician prior to participation -

Exclusion Criteria:

History of cardiovascular, respiratory, metabolic, neurological, or musculoskeletal disorders

Regular exposure to cold environments or cold water (cold-acclimatized individuals)

Use of medications that could affect thermoregulation or neuromuscular function

Any skin conditions that may be aggravated by cold water immersion

Inability to provide informed consent

Failure to pass pre-exposure medical examination by a study physician

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representattion
Study Population: The study population consists of healthy, active-duty male submariners from the Israeli Navy, aged 20 to 25 years. All participants were volunteers with no prior acclimatization to cold water or cold environments. Each participant underwent a medical screening by a qualified physician to confirm eligibility and provided written informed consent prior to participation. The cohort was selected to represent operationally relevant individuals likely to utilize Submarine Escape Immersion Equipment (SEIE) suits in real-world scenarios.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Core temperature | two hours
  Core temp. measured with telemetric pills

SECONDARY OUTCOMES:
Subjective cold sensation - | two hours
  Assessed using a standardized cold discomfort scale during immersion and raft sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Oren GABAY, MD, Principal Investigator — ISRAEL NAVAL MEDICAL INSTITUTE
Locations (1):
- Israel Naval Medical Institute, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
The raw, de-identified data collected during the study will be made available upon reasonable request. The dataset contains no personally identifiable information and includes only aggregated physiological and performance measurements. Data will be shared for academic, scientific, or regulatory purposes following review and approval by the principal investigator. Requests can be directed to the corresponding author.